CLINICAL TRIAL: NCT04947982
Title: Low Versus Standard Pressure Pneumoperitoneum in Laparoscopic Gynecological Surgery: A Randomized Controlled Trial
Brief Title: Low Versus Standard Pressure Pneumoperitoneum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, KG, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUGLA-4
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Gynecologic Surgery
MeSH Terms: interventions — Carbon Dioxide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): All laparoscopic surgical procedures were performed at 12 mmHg CO2 pressure throughout the surgery
- Study (Experimental): All laparoscopic surgical procedures were performed at 8 mmHg CO2 pressure throughout the surgery
  Interventions: Other: carbon dioxide

INTERVENTIONS:
Other: carbon dioxide — carbon dioxide insufflation pressure
  Arms: Study

SUMMARY:
The role of laparoscopy in gynecological and gyne-oncological surgery has dramatically increased over the past decades. Although laparoscopic procedure has several advantages over open surgery such as reduced blood loss, faster recovery earlier return to normal activities and work, however, postoperative pain and some hemodynamic changes sometimes discomforts the patients, lessening quality of life at postoperative period [1-3]. In clinical practice the majority of laparoscopic procedures are performed using standard pressure pneumoperitoneum (SPP, 12-15 mmHg) [1-3]. These noticeable adverse effects are associated with of creation of pneumoperitoneum with carbon dioxide (CO2) but it is requisite in all laparoscopic surgery for adequate visualization and operative manipulation.

The incidence of pain after gynecologic laparoscopies has been reported to vary from 35% to 63% [4,5]. A randomized controlled trial has demonstrated that there may be more intense pain and greater analgesia requirements in the immediate postoperative period after laparoscopic surgery than after laparotomy [6]. The origin of pain after laparoscopy is multifactorial and complex. It can be differentiated into abdominal pain and shoulder pain [7]. The precise causes for such pain are still obscure. Abdominal pain may be attributed to stretching of the abdominal cavity, and peritoneal irritation due to entrapment of dissolved CO2 [1-7]. Intraperitoneal acidosis, mucosal ischemia and compression of the splanchnic nerve as a consequence of the pneumoperitoneum may also be relevant factors [8,9]. On the other hand, shoulder pain is related to phrenic nerve and diaphragm irrigation due to residual CO2 in the subdiaphragmatic space [7-9].

In addition to pain, CO2 insufflation and a concomitant steep head-down (Trendelenburg, TP) position in surgical procedure also cause an increase in intra-abdominal pressure, which unfavorably affect patients homeostasis, inducing a significant change in the respiratory and cardiovascular system, lessening perfusion in abdominal organs and blood flow in the inferior vena cava, and posing an increased risk of thrombotic disease [10,11].

Low-pressure pneumoperitoneum (LPP, 7-10 mmHg) is recommended to minimize the adverse side effects associated with SPP [12]. There are several reports on the safety of low CO2 pneumoperitoneum pressure (LPP) in gynecological laparoscopic procedures however their trials have some limitations due to the small sample size, performed in only short laparoscopic procedures, and inadequate to assess the surgical impression of visualization [13-16]. Thus, further studies are still required.

Therefore, the purpose of this randomized controlled trial (RCT) is to assess the effect of LPP versus SPP on metabolic response, postoperative pain scores, surgical field visualization.

ELIGIBILITY:
Inclusion Criteria:

* Women underwent a total laparoscopic hysterectomy with or without additional surgery, such as salpingo-oophorectomy, salpingectomy, or pelvic and/or para-aortic lymphadenectomy

Exclusion Criteria:

* those who refused to give consent
* inability to understand the research questionnaire
* severe psychiatric or mental disorders
* American Society of Anesthesiologists (ASA) physical status classification > III
* conversion to laparotomy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Quality of postoperative recovery | at 24 hours after the surgical procedure (postoperative day [POD] 1)
  QoR-40 questionnaire scores. This questionnaire pertains to five dimensions of recovery: physical comfort (12 questions), emotional state (9 questions), physical independence (5 questions), psychological support (7 questions), and pain (7 questions). Each question carries 5 point Likert scale (none of the time, some of the time, usually, most of the time, and all of the time). The total score on the QoR-40 ranges from 40 (poorest possible recovery) to 200 (best possible recovery)

SECONDARY OUTCOMES:
Abdominal and shoulder pain intensities | The pain score were measured every 6 hours for 48 hours after surgery.
  Before starting the study, the participants will be instructed on how to assess their pain intensity using a visual analog scale (VAS; 0 cm = no pain, 10 cm = worst pain imaginable). To improve adherence to the protocol, participants will be asked to request analgesia without hesitation if the VAS pain score is > 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Education and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided